CLINICAL TRIAL: NCT05667350
Title: Exploration and Validation of a Diagnosis Model for Biliary Tract Cancer Based on Combined Liquid Biopsy in Peripheral Blood: A Multi-center Prospective Study
Brief Title: AssesSment of Early-deteCtion basEd oN liquiD Biopsy in Biliary Tract Cancer (ASCEND-BTC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Collaborators: Guangzhou Burning Rock Bioengineering Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Xiaoqing Jiang, Director, Eastern Hepatobiliary Surgery Hospital
Other Study IDs: RSCD2021021
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, white blood cells and fresh frozen tumor tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer arm: Baseline blood samples will be collected from participants newly diagnosed with biliary tract cancer.
  Interventions: Other: Blood drawing
- Benign disease arm: Baseline blood samples will be collected from participants newly diagnosed with benign biliary tract diseases.
  Interventions: Other: Blood drawing

INTERVENTIONS:
Other: Blood drawing — Blood drawing before anti-cancer therapy
  Groups: Cancer arm
Other: Blood drawing — Blood drawing before radical treatment
  Groups: Benign disease arm

SUMMARY:
ASCEND-BTC is a prospective, multi-center, observational study aimed at detecting early biliary tract cancer by combined assays of serum protein and cell-free DNA (cfDNA) methylation. The study will enroll approximately 492 participants diagnosed with biliary tract cancer and benign diseases.

ELIGIBILITY:
Inclusion Criteria for Cancer Arm Participants:

* Age 40-75 years at the day of consenting to the study.
* Able to provide a written informed consent
* Pathologically confirmed biliary tract cancers.
* No prior or ongoing anti-cancer therapy (local or systematic) prior to study blood draw.

Exclusion Criteria for Cancer Arm Participants:

* Pregnancy or lactating women.
* Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant.
* Recipients of blood transfusion within 7 days prior to study blood draw.
* Recipients of any anti-cancer therapy within 30 days prior to study blood draw, due to diseases other than cancers.
* With other known malignant tumors or multiple primary tumors.

Inclusion Criteria for Benign Arm Participants:

* Age 40-75 years at the day of consenting to the study.
* Able to provide a written informed consent.
* Confirmed diagnosis of benign biliary tract diseases.
* No prior radical treatment of the benign diseases prior to study blood draw.

Exclusion Criteria for Benign Arm Participants:

* Pregnancy or lactating women.
* Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant.
* Recipients of blood transfusion within 7 days prior to study blood draw.
* Recipients of any anti-cancer therapy within 30 days prior to study blood draw, due to diseases other than cancers.
* Confirmed diagnosis of malignancies or precancerous lesion.
* A history of malignant tumors.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from participating medical centers and assigned into two arms, including participants with new diagnosis of biliary tract cancer and benign biliary tract diseases.
Sampling Method: Non-Probability Sample
Enrollment: 492 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of the combined model in detection of biliary tract cancers. | 24 months

SECONDARY OUTCOMES:
The sensitivity and specificity of the combined model in detection of different subtypes of biliary tract cancers. | 24 months
The sensitivity and specificity of the combined model in detection of different stages of biliary tract cancers. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqing Jiang, MD/PhD, Principal Investigator — Eastern Hepatobiliary Surgery Hospital; Bin Li, MD/PhD, Principal Investigator — Eastern Hepatobiliary Surgery Hospital
Locations (2):
- China (2):
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality